CLINICAL TRIAL: NCT00156806
Title: Investigating the Therapeutic Effectiveness of Aloe Barbadensis in Reducing Cutaneous Side-Effects of Radiation Treatment for Breast Cancer.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AHS Cancer Control Alberta (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: PS-08-0006
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: Breast Cancer
Keywords: aloe; radiation dermatitis; radiation therapy
MeSH Terms: conditions — Breast Neoplasms; Radiodermatitis

INTERVENTIONS:
Procedure: Aloe barbadensis topical application in a moisturizing cream vehicle.

SUMMARY:
Breast cancer treatment often involved radiation to the breast. A side-effect of this treatment is skin redness, itching and burning. Some patients have quite severe reactions. Our current treatment for this is to avoid any soaps or other skin irritants and to use a moisturizing cream once all radiation is finished. Aloe vera is believed by many people to be useful for treatment of skin burns but this has never been proven in a randomized study. The aim of this study is to compare aloe vera gel versus plan gel versus the standard treatment to determine if there is any benefit. If there was a benefit of gel treatment over standard it could make radiation treatments more tolerable for cancer patients.

DETAILED DESCRIPTION:
BackgroundRadiation therapy is an important component of treatment for breast cancer, especially in the setting of breast conservation. Even though cancer patients who are receiving radiation treatments follow established hygiene and skin-care protocols they still experience differing degrees of cutaneous skin reactions and associated symptoms of dryness, itchiness, burning sensations, and pain.1-7 For some patients the side-effects associated with radiation therapy can become so severe serious consideration is given to discontinuing treatments. The treatments currently used for reducing cutaneous reactions and symptoms are very limited and often ineffective.5-7 Anti-inflammatories and steroid-based topical pharmaceutical agents are used sparingly due in part to research findings8 and potential harmful side-effects.7 This has left physicians and patients using a trial and error approach in seeking an alternative treatment that will help these patients cope with (and sometimes endure) the cutaneous radiation side-effects. Ongoing clinical experience and discussions with present and former radiation patients reveals that skin irritation, breakdown, pain and associated suffering are common side-effects that patients wish they did not have to experience. The lack of effective, efficient, non-pharmacological treatments for reducing symptoms associated with cutaneous skin reactions to radiation cancer therapy is problematic. Study Objectives the overall aim of the study is to determine if biologically active A. barbadensis is a therapeutic agent for reduction of cutaneous side effects women experience as a result of undergoing radiation therapy for breast cancer.The primary aim is to determine if there is a significant reduction or increase of cutaneous skin reactions using A. barbadensis on the irradiated skin of the breast or chest wall in comparison to following the standard CCI non-pharmacological treatment protocol and in comparison to using the moist inert vehicle gel on the irradiated site.The secondary aim is to explore if there is a reduction or increase in subjective symptoms at the irradiated site with the use of A. barbadensis in comparison to following the standard CCI 'best care' non-pharmacological treatment protocol and in comparison to using the moist inert vehicle gel on the irradiated site.MethodThis study is a single blind randomized controlled trial using a three Arm design. Analysis stratification is being conducted according to radiation technique, breast size, smoker vs. non-smoker, nutrition, protocol adherence, and prior chemotherapy. The control arm will treat the skin reaction as per standard CCI breast radiation protocol

ELIGIBILITY:
Inclusion Criteria:

* adult age women receiving 4500cGy or 5000cGy for non-metastatic breast cancer.
* tumor bed boost allowed.

Exclusion Criteria:

* patients with uncontrolled diabetes, uncontrolled eating disorder, acquired immunodeficiency syndrome, active lupus or scleroderma, a known allergy to pure aloe gel, a pre-study contact dermatitis to study creams.
* consenting procedures not completed prior to 10cGy of radiation therapy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 231
Dates: Start 2002-03; Primary Completion 2005-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Skin reaction severity.

SECONDARY OUTCOMES:
Symptom severity.

CONTACTS AND LOCATIONS:
Overall Officials: Donna L. Hoopfer, PhD, Principal Investigator — AHS Cancer Control Alberta
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada